CLINICAL TRIAL: NCT07134595
Title: A Multicenter Study Comparing Conventional Continuous Ambulatory Peritoneal Dialysis Prescription (C-CAPD) With Modified-CAPD (M-CAPD) Prescription in Delivering High Quality Goal-directed Peritoneal Dialysis in Children With End-stage Kidney Disease From Low-resource Settings: MaxED-OUT Trial
Brief Title: Comparing Conventional Continuous Ambulatory Peritoneal Dialysis Prescription (C-CAPD) With Modified-CAPD (M-CAPD) Prescription in Children With End-stage Kidney Disease From Low-resource Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Collaborators: University of the Philippines Manila - Philippine General Hospital (Other); Hospital Tuanku Jaafar, Seremban, Negeri Sembilan (Unknown); Dr. Soetomo General Hospital (Other Government); Pediatric Institute, Hospital Kuala Lumpur (Unknown)
Responsible Party: Principal Investigator, Sharon Teo, Consultant, National University Health System, Singapore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UPMREB 2024-0138-01
Record Dates: First submitted 2025-07-21; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Children on Chronic Peritoneal Dialysis
Keywords: M-CAPD; C-CAPD; ESKD; Children; Low-resource settings

STUDY DESIGN:
Intervention Model Description: A computer-generated random number will be assigned to patients to undergo either C-CAPD or M-CAPD therapy. After randomization, a 2-week run-in period will precede the assigned CAPD prescription. They will perform this assigned PD prescription for 2 consecutive months. After which, a 2-week wash-out period will be allowed before crossing over to either C-CAPD or M-CAPD. The total intervention time is 12 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- C-CAPD therapy (Active Comparator): The prescription for the C-CAPD therapy is as follows:
  1. PD solution containing 1.5%, 2.5% dextrose (or its equivalent, for example, 2.3%), 4.25%.
  2. Full fill volume computed as 1100-1400 ml/m2 as described by Fischbach et al. [19],
  3. Day-time and night-time dwell time ranging from 3 to 6 hours
  4. Two to 3-daytime exchanges with or without night exchange
  5. 8 to 10 hours of overnight dwell
  Interventions: Other: C-CAPD Prescription; Other: M-CAPD Prescription
- M-CAPD Therapy (Experimental): The prescription for the M-CAPD therapy is the C-CAPD with an additional 1 to 2 short, low-volume, 15 to 30-minute dwells per exchange before instilling the computed full dwell volume.
  Interventions: Other: C-CAPD Prescription; Other: M-CAPD Prescription

INTERVENTIONS:
Other: C-CAPD Prescription — The prescription for the M-CAPD therapy is the C-CAPD with an additional 1 to 2 short, low-volume, 15 to 30-minute dwells per exchange before instilling the computed full dwell volume.
  Other Names: M-CAPD Prescription
Other: M-CAPD Prescription — The prescription for the M-CAPD therapy is the C-CAPD with an additional 1 to 2 short, low-volume, 15 to 30-minute dwells per exchange before instilling the computed full dwell volume.

SUMMARY:
This study aims to compare modified CAPD (M-CAPD) and conventional CAPD (C-CAPD) in terms of delivering high-quality, goal-directed PD as well as avoiding resource wastage in prevalent ESKD patients aged 2 to ≤18 years using a randomized cross-over study design for one year.

This study hypothesizes that M-CAPD will have better ultrafiltration and solute clearance than C-CAPD.

Specific objectives

1. To determine the ultrafiltration efficiency by measuring the following:

   1. Clinical parameters: blood pressure, weight, evidence of fluid overload by the presence of edema, abnormal heart sounds (S3 gallop), lung crackles or rales, increased heart rate (tachycardia), rapid breathing (tachypnea),
   2. Change in the number of blood pressure medications before and after the intervention,
   3. Absolute and relative fluid overload using bioimpedance analyzer (BIA),
   4. Mean daily ultrafiltration (UF) or Total 24-h UF,
   5. Residual kidney function: 24-hour urine output,
   6. Glucose exposure
2. To determine the solute clearance adequacy by measuring the following:

   1. Serum sodium, chloride, potassium, bicarbonate, serum albumin, calcium, and hemoglobin,
   2. Phosphate clearance
   3. Renal and peritoneal Kt/Vurea
   4. Normalized protein catabolic rate (nPCR)
3. To measure caregiver burden using a Paediatric Renal Caregiver Burden Scale (PR-CBS).

DETAILED DESCRIPTION:
Background and Rationale Peritoneal dialysis (PD) is the primary kidney replacement therapy (KRT) for children with end-stage kidney disease (ESKD), particularly in low-resource settings. In these settings, continuous ambulatory peritoneal dialysis (CAPD) is more accessible than automated PD (APD) or hemodialysis due to the lack of power and expensive machinery.

However, standard CAPD regimens can lead to significant wastage of PD fluid. For example, using standard 2-liter bags, children often use only a portion of each bag, discarding the rest. Additionally, fixed-volume, fixed-dwell CAPD is often suboptimal for solute clearance and ultrafiltration, particularly in patients with different peritoneal membrane transport types.

Adapted APD (aAPD), pioneered by Fischbach et al., offers a better solution by combining short, low-volume exchanges with longer, high-volume ones to improve ultrafiltration and solute clearance. This study proposes a Modified CAPD (M-CAPD) that incorporates the principles of aAPD but adapted for manual (non-automated) settings.

Rationale No existing studies have applied the aAPD approach to CAPD in children or adults. This study addresses both clinical effectiveness and resource optimization in PD for children in Southeast Asia.

General Objective

To compare Modified CAPD (M-CAPD) and Conventional CAPD (C-CAPD) in terms of:

* Clinical outcomes (ultrafiltration, solute clearance),
* Resource utilization (waste reduction),
* Caregiver burden. Specific Objectives

  1. Ultrafiltration Efficiency i. Clinical parameters: BP, weight, edema, S3 gallop, lung crackles, tachycardia, tachypnea.

     ii. Number of antihypertensive medications. iii. Bioimpedance analysis (BIA). iv. Total 24-hour UF and residual urine output. v. Glucose exposure per day.
  2. Solute Clearance Adequacy i. Serum electrolytes (Na, Cl, K, HCO₃-, Ca), albumin, hemoglobin. ii. Phosphate clearance. iii. Renal and peritoneal Kt/V. iv. Normalized protein catabolic rate (nPCR).
  3. Caregiver Burden i. Measured using Pediatric Renal Caregiver Burden Scale (PR-CBS). Study Design
* Design: Prospective, multicenter, randomized cross-over trial.
* Duration: 12 weeks of active intervention per participant.
* Setting: Pediatric dialysis centers in the Philippines, Malaysia, and Indonesia.
* Run-in Period: 2 weeks
* Intervention Phases: Each participant undergoes both C-CAPD and M-CAPD for 8 weeks total (2 months per arm), with a 2-week washout in between.
* Randomization: Computer-generated random number assignment. Sample Size
* Assuming high correlation (r=0.95), 26 patients at PGH are sufficient (13 per arm). Total across centers: 44 children aged 2 to ≤18 years.

Intervention Details Conventional CAPD (C-CAPD)

* PD solutions: 1.5%, 2.5%, 4.25% dextrose
* Fill volume: 1100-1400 mL/m²
* 3-4 exchanges per day
* Day and night dwell times: 3-6 hours (day), 8-10 hours (night) Modified CAPD (M-CAPD)
* Follows C-CAPD with addition of 1-2 short, low-volume (15-30 min) exchanges before full-volume dwell.
* Short dwell volume comes from remaining solution in the 2L bag. Monitoring and Follow-Up
* Every 2 weeks (remote or in-person)
* Monitored parameters: BP, HR, weight, edema, UF, urine output
* Data collection notebook maintained by patient/caregiver Adverse Events Monitoring

Includes:

* Exit site infection
* Peritonitis
* Hypertension or fluid overload
* Dehydration (over-UF)
* Hyperglycemia
* Hospitalization
* Withdrawal criteria detailed Outcome Measures and Data Collection Timepoints: Baseline, post-randomization (6 weeks), post-crossover (12 weeks)

Data Collected:

* Physical exam, vital signs, UF/urine output
* Lab values: electrolytes, albumin, hemoglobin, FBS
* Bioimpedance analysis
* Kt/V, nPCR
* PR-CBS for caregiver burden Data Analysis Plan
* Descriptive statistics: for demographics and baseline data
* Paired t-tests: for continuous outcomes
* McNemar's test: for categorical outcomes (e.g., edema)
* Outcomes compared within subjects (cross-over design) Ethical Considerations
* Guidelines followed: Declaration of Helsinki, ISO 14155:2011, Good Clinical Practice, Philippine Data Privacy Act (2012)
* Ethics approval: To be obtained from institutional ethics boards
* Informed consent: Required from caregivers; assent from children ≥6 years Risks
* Minor discomfort from added blood draws
* No added infection risk from M-CAPD as procedure remains closed
* Risks managed with prompt clinical support and compensation Benefits
* Improved PD efficiency and fluid management
* Reduced glucose exposure and complications
* Less wastage of PD fluid
* Cost savings for families
* Enhanced caregiver education and burden reduction
* Potential improvement in health-related quality of life Compensation
* Covers: PD supplies, lab tests, transport, meals
* Provides treatment for study-related injuries
* Free antibiotics for PD-related infections Privacy and Confidentiality
* Strict adherence to data protection guidelines
* Anonymized data with unique identifiers
* Secure physical and digital storage
* Data access restricted to PI and trained assistant
* All data deleted within 2 years of study conclusion Dissemination Plan
* Results to be shared with physicians, caregivers, and published in peer-reviewed journals
* All data anonymized in reports Intellectual Property and Legal Compliance
* Pre-existing IP remains with originator
* Jointly generated IP to be co-owned
* Philippine laws and UP policies govern research conduct Vulnerable Populations
* Pediatric patients with ESKD from lower socioeconomic backgrounds
* Extra care in informed consent and ethical oversight

ELIGIBILITY:
Inclusion Criteria:

* CKD 5D who have been on peritoneal dialysis for at least three months.

Exclusion Criteria:

1. Patients with BSA of ≥1.5 m2,
2. Evidence of mechanical causes of low ultrafiltration capacity (hernia, peri-catheter, or genital leaks, pleuroperitoneal communication),
3. Peritoneal membrane failure (encapsulating peritoneal sclerosis),
4. Recent episode of peritonitis (within two months)
5. Those who have been on hemodialysis before switching to PD in the last three weeks.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Ultrafiltration efficiency | 12 weeks
  Ultrafiltration (UF): Assessed clinically through blood pressure, presence of edema or crackles, reduced need for antihypertensive medications, residual kidney function, and mean daily UF.
The solute clearance adequacy | 12 weeks
  Toxin Removal: Evaluated by comparing pre- and post-intervention levels of electrolytes and urea clearance, calculated using the Kt/V formula.

SECONDARY OUTCOMES:
To measure caregiver burden | 12 weeks
  Caregiver burden will be measured by using a Paediatric Renal Caregiver Burden Scale (PR-CBS) Using the Caregiver Burden Scale (1-5, with higher scores indicating greater burden), we will assess whether the additional exchange is perceived as an increased burden or a relief, particularly if clinical improvements in the child are observed.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Kim Yap, Professor, Principal Investigator — National University Health System, Singapore
Locations (1):
- Philippine General Hospital, Manila, Ermita, Philippines

IPD SHARING:
Plan to Share IPD: No